CLINICAL TRIAL: NCT07181824
Title: VAP Incidence and Adequation to SRLF 2017 Diagnostic Among an Intensive Care Medicine Service for the Period 2022 à 2024
Acronym: PAVM-RéaCHSF
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Other Study IDs: 2025/0025
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Pneumonia Ventilator Associated
Keywords: Ventilatory associated pneumonia; VAP; Intensive Care medicine; Mechanical ventilation; Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- VAP suspicion: Adult patients (>18 years) under mechanical ventilation for >48 hours and with a positive respiratory sample
  Interventions: Other: Diagnostic tedst

INTERVENTIONS:
Other: Diagnostic tedst — * Radiologic signs: 2 consecutive thorax x-ray with new onset pneumonia AND
  * One of the following criteria
    * Fever >38,3°C without any other cause
    * Leucocytes < 4000/mm3 or ≥ 12000 /mm3
  * AND at least two of the following
    * Purulent secretions
    * Cough or dyspnoea
    * Desaturation or increase in FiO2 (+20%)

SUMMARY:
The goal of this observational study is to to analyze respiratory samples performed in mechanically ventilated ICU patients and to assess whether the SRLF criteria for defining VAP were respected among patients admited to the Intensive care medicine at a regional hospital en France

DETAILED DESCRIPTION:
Ventilator-associated pneumonia (VAP) is a lung infection that occurs after more than 48 hours of mechanical ventilation. It is of particular interest because it affects between 5-40% of ICU patients depending on the study and diagnostic criteria, with a relatively low attributable mortality (around 10%), but with increased morbidity, notably in terms of the duration of mechanical ventilation and ICU length of stay. In addition, it is the leading cause of nosocomial infection in the ICU, accounting for up to 25% of antibiotic use for hospital-acquired infections.

The diagnosis of VAP is based on clinico-radiological criteria: the appearance or worsening of a radiological pulmonary infiltrate, an inflammatory syndrome, the appearance of secretions, increased oxygen dependency and/or worsening of shock, confirmed by a positive respiratory sample.

The diagnostic challenge lies in the fact that the signs and symptoms are not pathognomonic of VAP and may be common to other conditions. On the other hand, patients may be colonized by pathogens without actually having VAP.

For this reason, scientific societies propose criteria to better target patients for whom a respiratory sample should be taken and antibiotic therapy initiated.

In 2017, the French Society of Intensive Care Medicine (SRLF) and the French Society of Anaesthesia and Intensive Care (SFAR) published recommendations on ICU-associated pneumonia, with some minor variations compared with the 2005 ATS/IDSA criteria.

Our study aims to analyze respiratory samples performed in mechanically ventilated ICU patients and to assess whether the SRLF criteria for defining VAP were respected.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years
* Hospitalization in Intensive care unit for the period between 01/01/2022 and 31/12/2024
* Intubation and mechanical ventilation for > 48h
* Positive respiratory sample

Exclusion Criteria:

* Decision of therapeutic limitation
* Organ donors
* Patient refuse to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population includes all patients admitted to the intensive care unit for the selected period, under mechanical ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
SRLF VAP criteria | at day 0
  Describe whether the respiratory samples obtained from ICU patients after >48 hours of mechanical ventilation for suspected VAP met, or did not meet, the 2017 SRLF diagnostic criteria

SECONDARY OUTCOMES:
microbial ecology in the ICU of CHSF | at day 0
  Prevalence of MDR in the respiratory samples
antibiotic consumption generated by VAP | at day 0
  To evaluate antibiotic consuming related to VAP episodes to the total antibiotic consuming in the Intensive care unit
morbidity and mortality associated with VAP | at day 0
  Mortality and mechanical ventilation duration among patients diagnosed of VAP
duration of antibiotic therapy for a VAP episode | at day 0
  Duration of antibiotherapy among patients with VAP
characteristics of the initial antibiotic therapy | at day 0
  Number and class of antibiotics of the initial antibiotic therapy
Evaluate the adequacy of the initial antibiotic therapy | at day 0
  Adequation of the initial therapy compared to the definitive therapy: maintain, increase or reduce the spectrum or number of antibiotics

CONTACTS AND LOCATIONS:
Overall Officials: Luis ENSENYAT MARTIN, MD, Principal Investigator — Centre Hospitalier Sud Francilien; Abdoul DINE, Study Director — Centre Hospitalier Sud Francilien
Locations (1):
- Centre Hospitalier Sud Francilien, Corbeil-Essonnes, France, France

IPD SHARING:
Plan to Share IPD: No